CLINICAL TRIAL: NCT04226196
Title: Rotational Stability of a Hydrophobic Acrylic Plate Haptic Intraocular Lens Using a Capsular Tension Ring - An Intraindividual Comparative Study
Acronym: ConTRol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Ao. Univ. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ConTRol
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Intraocular Lens Rotation; Capsular Tension Ring
Keywords: Intraocular lens rotation; capsular tension ring; postoperative tilt & decentration

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator will be masked to which axis the IOL will be implanted until a sealed envelope will be opened in the operating theater.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Axis 0 (Experimental): IOL Implantation at the 0 +/- 10 degrees axis
  Interventions: Device: Implantation of an intraocular lens
- Axis 45 (Experimental): IOL Implantation at the 45 +/- 10 degrees axis
  Interventions: Device: Implantation of an intraocular lens
- Axis 90 (Experimental): IOL Implantation at the 90 +/- 10 degrees axis
  Interventions: Device: Implantation of an intraocular lens
- Axis 135 (Experimental): IOL Implantation at the 135 +/- 10 degrees axis
  Interventions: Device: Implantation of an intraocular lens

INTERVENTIONS:
Device: Implantation of an intraocular lens — Implantation of an intraocular lens Zeiss 409 MP into the capsular bag using an injector, after removing of the human crystalline lens.

SUMMARY:
The present study should investigate the influence of a capsular tension ring on postoperative rotational stability of a plate haptic hydrophilic acrylic intraocular lens. All patients will be operated on both eyes in one occasion. Both eyes receive a Zeiss 409MP plate haptic intraocular lens, while only on eye receives an additional capsular tension ring. Follow up visits take place 1 hour, 1 week, 1 month and 4 to 7 months after surgery. At the follow up visits, the actual IOL axis will be determined by retroillumination photography. IOL centration and tilt will be determined by anterior segment SS-OCT Casia II. IOLs will be implanted in 4 different axis 0 +/- 10 degrees, 45 +/- 10 degrees, 90 +/- 10 degrees, 135 +/- 10 degrees. IOL rotation, decentration and tilt then will be compared intraindividually.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract necessitating phacoemulsification extraction and posterior IOL implantation
* Need for spherical IOL correction between +0.00 and +32.00 D
* Pupil dilation of ≥ 7.0 mm
* Age 45 to 95

Exclusion Criteria:

* Corneal abnormality (Corneal scaring)
* Preceding ocular surgery or trauma
* Uncontrolled glaucoma
* Proliferative diabetic retinopathy
* Iris neovascularization
* History of uveitis/iritis
* Microphthalmus
* Recurrent intraocular inflammation of unknown etiology Uncontrolled systemic or ocular disease
* Pregnancy
* Lactation

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Change of axial intraocular lens position | 7 months
  Change in axis position of an intraocular lens Zeiss 409 MP from end of surgery (baseline axis) to 1 hour, 1 week, 1 month and 4-7 months (end of study visit). The change in axis position will be evaluated with respect to the baseline measurement at the end of surgery. Differences in axis position will be described as rotation in degrees (0 to 360°)

SECONDARY OUTCOMES:
Decentration | 7 months
  Decentration of the intraocular lens will be measured with the Casia 2 OCT. Decentration will be described as "Decentration in millimeter"
Tilt | 7 months
  Tilt of the intraocular lens will be measured with the Casia 2 OCT. Tilt will be described as "Tilt in degrees at a certain axis"
Anterior chamber depth | 7 months
  The anterior chamber depth (Axial position of the IOL) of the intraocular lens will be measured with the Casia 2 OCT after 1 month. The anterior chamber depth will be measured in millimeter
Best corrected visual acuity (BCVA) | 7 months
  BCVA will be measured at 1 week, 1 month and 4 to 7 months. The BCVA will be described as the minimum angle of resolution (logMar)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna Allgemeines Krankenhaus, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided